CLINICAL TRIAL: NCT03892460
Title: Novel Transitional Rehabilitation Care in Coronary Artery Bypass Graft (CABG) Patients
Brief Title: Transitional Rehabilitation in CABG Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Michael J. Toth, Ph.D., Professor of Medicine, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-0413
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Results first posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Coronary Artery Disease; Coronary Artery Bypass Graft Surgery
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental): Neuromuscular electrical stimulation
  Interventions: Device: neuromuscular electrical stimulation
- Control (No Intervention): No treatment control

INTERVENTIONS:
Device: neuromuscular electrical stimulation — bilateral quadriceps exercise with neuromuscular electrical stimulation
  Arms: Treatment

SUMMARY:
The goal of this research study is to understand whether an at-home exercise program started soon after CABG surgery, and continuing for 4 weeks following discharge from the hospital, can preserve or improve physical function.

DETAILED DESCRIPTION:
Coronary artery bypass graft (CABG) surgery is a common surgical procedures and an important treatment option for coronary artery disease. The post-surgery period of rest and recovery is associated with cardiorespiratory and skeletal muscle deconditioning. The goal of this research study is to understand whether an at-home exercise program started soon after CABG surgery, and continuing for 4 weeks following discharge from the hospital, can serve as a bridge between surgery and the start of cardiac rehabilitation to preserve or improve physical function. Volunteers will be randomly assigned to receive neuromuscular electrical stimulation (NMES) of their quadriceps muscles or not to receive NMES (control group). Volunteers will be evaluated prior to CABG, upon discharge and 4 weeks Post-CABG surgery. Assessments will include measurements of physical function by the Short Physical Performance Battery, 6 min walk tests and body composition analysis, as well as assessment of subjective physical functional capacity and quality of life using the Medical Outcomes Short form 36. Additionally, accelerometry will be used to monitor weight-bearing physical activity during the 4 week treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* 50-80 yrs of age
* ambulatory
* scheduled for coronary artery bypass graft surgery
* able to provide informed consent

Exclusion Criteria:

* rheumatoid arthritis or other inflammatory/autoimmune disease
* cancer, excluding non-melanoma skin cancer
* exercise limiting peripheral vascular disease
* neuromuscular disease or neuromuscular dysfunction associated with cerebrovascular event
* body mass index >38 kg/m2
* valvular heart disease not corrected surgically
* lower extremity blood clot or implantable cardioverter-defibrillator

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2019-10-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont College of Medicine, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rengo JL, Savage PD, Hirashima F, Leavitt BJ, Ades PA, Toth MJ. Improvement in Physical Function After Coronary Artery Bypass Graft Surgery Using a Novel Rehabilitation Intervention: A RANDOMIZED CONTROLLED TRIAL. J Cardiopulm Rehabil Prev. 2021 Nov 1;41(6):413-418. doi: 10.1097/HCR.0000000000000576. PMID 33512980

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 30 | 24
Randomization | 25 | 20
Completed | 18 | 19
Not Completed | 12 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 30 | 24 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (5.9) | 66.5 (7.1) | 65.7 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 27 | 21 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 29 | 24 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 28 | 24 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 24 | 54

OUTCOME MEASURES:

1. Primary Outcome: Short Physical Performance Battery
Description: Short Physical Performance Battery is composed of three tasks assessing balance, gait speed, and ability to stand from a chair. Units on a scale for each domain range from of 0-4 for a total score of 0 to 12, with a higher score indicating better physical function.
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 18 | 19
units on a scale
  Discharge | 7.33 (0.55) | 8.00 (0.54)
  4-weeks post-discharge | 11.44 (0.22) | 10.90 (0.21)

2. Secondary Outcome: 6 Minute Walk Distance
Description: 6 MW was developed to assess cardiopulmonary fitness in patients with lung and cardiac disease, and has been validated in cardiac surgery patients. It assesses the distance that a patient can walk in 6 minutes time around a standard course.
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: meters
Arm/Group | Treatment | Control
Number analyzed (Participants) | 18 | 19
meters
  Discharge | 216 (22) | 238 (21)
  4-weeks post-discharge | 482 (21) | 431 (20)

3. Secondary Outcome: Medical Outcomes Short Form 36 - Physical Function
Description: The Medical Outcomes Short Form 36 is a questionnaire that assesses self-reported health and physical functional status. There are 36 questions that reflect eight sub-domains of health included in this questionnaire. Scores for each domain represent weighted sums of the questions in each sub-domain. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. This sub-domain focused on limitations in physical function due to health problems. Lower scores represent more physical function disability, while higher scores represent less disability.
Time Frame: Hospital discharge and 4-weeks post-discharge
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 18 | 19
units on a scale
  Discharge | 40 (7) | 33 (7)
  4-weeks post-discharge | 70 (5) | 58 (5)

4. Secondary Outcome: Medical Outcome Short Form 36 - Role Physical
Description: The Medical Outcomes Short Form 36 is a questionnaire that assesses self-reported health and physical functional status. There are 36 questions that reflect eight sub-domains of health included in this questionnaire. Scores for each domain represent weighted sums of the questions in each sub-domain. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. This sub-domain focused on limitations in usual role activities because of physical health problems. Lower scores represent more disability, while higher scores represent less disability.
Time Frame: Hospital discharge and 4-weeks post-discharge
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 18 | 19
units on a scale
  Discharge | 26 (10) | 21 (9)
  4-weeks post-discharge | 19 (8) | 18 (7)

5. Secondary Outcome: Medical Outcomes Short Form 36 - Bodily Pain
Description: The Medical Outcomes Short Form 36 is a questionnaire that assesses self-reported health and physical functional status. There are 36 questions that reflect eight sub-domains of health included in this questionnaire. Scores for each domain represent weighted sums of the questions in each sub-domain. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. This sub-domain focused on bodily pain. Lower scores represent more pain, while higher scores represent less pain.
Time Frame: Hospital discharge and 4-week post-discharge
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 18 | 19
units on a scale
  Discharge | 31 (4) | 28 (4)
  4-weeks post-discharge | 28 (3) | 27 (3)

6. Secondary Outcome: Medical Outcomes Short Form 36 - General Health
Description: The Medical Outcomes Short Form 36 is a questionnaire that assesses self-reported health and physical functional status. There are 36 questions that reflect eight sub-domains of health included in this questionnaire. Scores for each domain represent weighted sums of the questions in each sub-domain. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. This sub-domain focused on self-reported general health. Lower scores represent worse health, while higher scores represent better health.
Time Frame: Hospital discharge and 4-week post-discharge
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 18 | 19
units on a scale
  Discharge | 71 (4) | 63 (4)
  4-weeks post-discharge | 81 (3) | 72 (3)

7. Secondary Outcome: Medical Outcomes Short Form 36 - Vitality
Description: The Medical Outcomes Short Form 36 is a questionnaire that assesses self-reported health and physical functional status. There are 36 questions that reflect eight sub-domains of health included in this questionnaire. Scores for each domain represent weighted sums of the questions in each sub-domain. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. This sub-domain focused on vitality (energy and fatigue). Lower scores represent less vitality, while higher scores represent more vitality.
Time Frame: Hospital discharge and 4-weeks post-discharge
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 18 | 19
units on a scale
  Discharge | 55 (5) | 53 (5)
  4-weeks post-discharge | 55 (4) | 51 (3)

8. Secondary Outcome: Medical Outcomes Short Form 36 - Social Function
Description: The Medical Outcomes Short Form 36 is a questionnaire that assesses self-reported health and physical functional status. There are 36 questions that reflect eight sub-domains of health included in this questionnaire. Scores for each domain represent weighted sums of the questions in each sub-domain. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. This sub-domain focuses on limitations in social activities because of physical or emotional problems. Lower scores represent more more limitations, while higher scores represent less lmitations.
Time Frame: Hospital discharge and 4-weeks post-discharge
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 18 | 19
units on a scale
  Discharge | 74 (7) | 63 (7)
  4-week post-discharge | 76 (6) | 72 (5)

9. Secondary Outcome: Medical Outcomes Short Form 36 - Role Emotional
Description: The Medical Outcomes Short Form 36 is a questionnaire that assesses self-reported health and physical functional status. There are 36 questions that reflect eight sub-domains of health included in this questionnaire. Scores for each domain represent weighted sums of the questions in each sub-domain. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. This sub-domain focuses on limitations in usual role activities because of emotional problems. Lower scores represent more limitations, while higher scores represent less limitations.
Time Frame: Hospital discharge and 4-week discharge
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 18 | 19
units on a scale
  Discharge | 65 (11) | 54 (11)
  4-week post-discharge | 72 (10) | 51 (9)

10. Secondary Outcome: Medical Outcomes Short Form 36
Description: The Medical Outcomes Short Form 36 is a questionnaire that assesses self-reported health and physical functional status. There are 36 questions that reflect eight sub-domains of health included in this questionnaire. Scores for each domain represent weighted sums of the questions in each sub-domain. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. This measure represents the total computed score across all sub-domains. Lower scores represent worse overall health, while higher scores represent better health.
Time Frame: Hospital discharge and 4-week post-discharge
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 18 | 19
units on a scale
  Discharge | 77 (4) | 74 (4)
  4-week post-discharge | 86 (4) | 78 (3)

11. Secondary Outcome: Physical Activity
Description: Physical activity was measured throughout the intervention in control and treatment groups and data. Data were analyzed by regression analysis to obtain the best fit line for the data and to compute a slope of the change in step count with day post-discharge to examine whether groups differed in their rate of recovery of weight-bearing activity (ie, walking).
Time Frame: Daily from discharge to 4-week post-discharge evaluation
Measure: Number; unit: step counts per day
Arm/Group | Treatment | Control
Number analyzed (Participants) | 18 | 19
step counts per day | 125.6 | 109.6

ADVERSE EVENTS:
Time Frame: 1-month post-surgery
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/24
Other Adverse Events (participants affected / at risk) | 1/30 | 0/24
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=30) | Control (N=24)
Pleuritic chest pain (Cardiac disorders) | 1 (30) | 0 (0) — Pleuritic chest pain during functional stesting

LIMITATIONS AND CAVEATS:
First, patients were not blinded to treatment status because NMES elicits skeletal muscle contraction and any sham treatment would not. Second, study personnel were not blinded, as resources were insufficient for unblinded and blinded personnel. Third, we did not analyze data using an intent-to-treat approach. Fourth, our study included few women. Finally, our study is limited to the strict inclusion/exclusion criteria and studies in larger cohorts are required to assess external validity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-17): https://cdn.clinicaltrials.gov/large-docs/60/NCT03892460/Prot_SAP_000.pdf